CLINICAL TRIAL: NCT07251452
Title: Effectiveness of a Dual Program of Physical Activity and Cognitive Intervention for Improving Sleep and Quality of Life in Older Adults.
Brief Title: Effectiveness of a Dual Program for Improving Sleep in Older Adults.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Laura Pilar de Paz Montón, Predoctoral researcher, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gerontology-sleep
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Sleep; Gerontology; Physical Therapy; Cognitive
Keywords: quality of life; sleep; physical activity; cognitive intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Talks are given on health education topics that are not related to the intervention to the participants.
  Interventions: Behavioral: Control
- Otago programme (Experimental): a physical activity intervention is applied to the participants.
  Interventions: Behavioral: Otago programme
- Otago programme + Cognitift (Experimental): a physical activity and cognitive training intervention is applied to the participants.
  Interventions: Behavioral: Otago programme + Cognifit

INTERVENTIONS:
Behavioral: Otago programme — Otago physical activity program adapted to elderly people
  Arms: Otago programme
Behavioral: Otago programme + Cognifit — Otago physical activity program adapted for seniors and cognitive training with the Cognifit app for smartphones or tablets.
  Arms: Otago programme + Cognitift
Behavioral: Control — Talks about topics of interest in health sciences not related to sleep
  Arms: Control

SUMMARY:
The present clinical trial aims to test whether a dual program of physical activity and cognitive training improves sleep and quality of life in people over 65 years of age.

DETAILED DESCRIPTION:
The intervention is being carried out in different day centers and co-housing centers in Toledo, Spain, where participants were recruited. A three-arm study was also conducted: a control group that received talks on health topics; a physical activity intervention group that followed the Otago physical activity program, tailored to; and a physical activity and cognitive training intervention group that used a mobile app known as Cognifit to develop the cognitive intervention.

ELIGIBILITY:
Inclusion Criteria:

* know how to use smartphones.
* have the ability to perform physical activity.

Exclusion Criteria:

* be under 65 years of age.
* suffer from serious pathologies that prevent the intervention from being carried out.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Sleep | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  Latency, sleep efficiency, number of awakenings during the night will be measured by actigraphy.
  The Pittsburgh Sleep Quality Index (PSQI) questionnaire will be used to asees objetive sleep quality and patterns in adults. It consists of 19 self-reported items. The 9 self-reported items of the PSQI generate seven component scores (with subscales ranging from 0 to 3): sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. The sum of these seven component scores produces an overall subjective sleep quality score (ranging from 0 to 21). Higher scores indicate poorer subjective sleep quality.

SECONDARY OUTCOMES:
Quality of life in older people | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  European Quality of Life 5 Dimensions (EQ-5D) will be used. Maximum score: 100, representing "best possible health." Minimum score: 0, representing "worst possible health."
Cognitive assessment and training | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  The CogniFit® computerized battery for smart devices is used for neurocognitive assessment and training of various cognitive functions, such as memory, attention, planning, processing speed, and cognitive flexibility. The CogniFit® neurocognitive assessment uses a series of interactive tasks and exercises to measure the status of different cognitive domains, providing detailed quantitative and graphical results that allow for the identification of strengths and areas for improvement. It has been previously validated in older adults, demonstrating good internal consistency (Cronbach's alpha = 0.85-0.88) and test-retest reliability (r = 0.69-0.92). The neurological assessment provides an overall score expressed in normative scores compared to similar populations, facilitating its interpretation in both clinical and research contexts. In addition, it offers cognitive training exercises.
Sociodemographic variables | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  Questionnaire on sociodemographic variables of own elaboration will be used for the collection of sociodemographic, anthropometric and health and drug-related data.
Degree of independence of older people in performing Basic Activities of Daily Living (BADLs) | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  The Katz Index, will be used to assess the level of independence of older adults in performing Basic Activities of Daily Living (BADLs). This instrument measures functional capacity in essential daily living tasks, providing an objective view of the level of dependence or autonomy of the person being evaluated. The index assesses six basic functions: bathing, dressing, toileting, mobility, continence, and feeding. (6) points: Independent in all activities. (0) points: Dependent in all activities.
Functional capacity in Instrumental Activities of Daily Living | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  The Lawton and Brody scale will be used to assess functional capacity in Instrumental Activities of Daily Living (IADLs), which are more complex tasks than basic activities and require more advanced cognitive and physical skills.
  0 points: Total dependence. 8 points: Total independence (for women, and 5 for men).
Level of social support and social network of older adults | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  The Lubben Social Network Scale (LSCS) will be used to assess the level of social support and social network of older adults. It consists of six items scored on a 0-to-5 Likert scale. Higher scores reflect larger social networks and greater availability of social support. Conversely, scores below indicate a high risk of social isolation.
Depression | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2 (8 weeks after the end of the intervention).
  Yesavage Geriatric Depression Scale will be used. Consists of 15 dichotomous (yes/no) questions, in which each item is scored 0 or 1 depending on the response.
  0-5 points: Normal. 6-9 points: Mild depression. > 10 points: Established depression.
Mobility | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2, 8 weeks after the end of the intervention.
  The Timed Up and Go (TUG) test will be used to assess balance, mobility, and fall risk in older adults. The test involves recording the time it takes a person to perform the following tasks: stand up from a chair with armrests, walk a distance of 3 meters marked on the floor, turn around, return to the chair, and sit down again. The total time is measured in seconds using a stopwatch. According to the standards, a time of less than 10 seconds indicates excellent mobility, while times greater than 20 seconds suggest limited mobility and a higher risk of falls.
Memory | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2, 8 weeks after the end of the intervention.
  The Memory Failures of Everyday (MFE) questionnaire will be used to assess everyday memory lapses. It consists of 28 items and is answered using a three-point Likert scale (Montejo et al. version) ranging from 'never in the last three months' to 'more than once a day'. Lower scores indicate fewer lapses, while higher scores indicate more lapses.
Cognitive disorders | Pre intervention T0 (one week before intervention started), post intervention T1 (after 12 weeks of intervention) and follow up T2, 8 weeks after the end of the intervention.
  Lobo Mini-Mental State Examination (36-item version) will be used to assess cognitive impairment associated with neurodegenerative diseases. It consists of several items that evaluate five cognitive domains: memory, orientation, attention span, calculation, concentration, and language. In geriatric patients over 65 years of age, scores below 23 are considered indicative of cognitive impairment; in patients under 65 years of age, scores of 27 or below are considered indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy and Nursing, Arms Factory, Toledo, 45071 Spain, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No